CLINICAL TRIAL: NCT00680485
Title: A Three Part Study in Healthy Adult Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of Repeat Escalating Oral Doses of GSK580416; the Safety, Tolerability, and Pharmacokinetics of GSK580416 Following a Loading Dose Regimen; and the Effect of Ketoconazole on the Pharmacokinetics of GSK580416
Brief Title: Evaluation of the Safety, Tolerability and Pharmacokinetics of Repeat Oral Doses of GSK580416
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OPS108221
Record Dates: First submitted 2008-04-14; First posted 2008-05-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Bacterial Infection; Infections, Bacterial
Keywords: GSK580416; ketoconazole interaction; pleuromutilin; oral dose
MeSH Terms: conditions — Bacterial Infections | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK580416 oral tablets (250 mg) Ketoconazole oral tablets (200 mg)

SUMMARY:
This study will evaluate the safety, tolerability and exposure of repeat escalating oral doses, a loading dose/maintenance dose regimen of GSK580416 and when co administered with ketoconazole, a PGP/CYP3A4 inhibitor.

DETAILED DESCRIPTION:
A three part study in healthy adult subjects to evaluate the safety, tolerability and pharmacokinetics of repeat escalating oral doses of GSK580416; the safety, tolerability, and pharmacokinetics of GSK580416 following a loading dose regimen; and the effect of ketoconazole on the pharmacokinetics of GSK580416

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (as determined by medical evaluation including history, physical exam, vital signs, laboratory tests, and cardiac monitoring)
* Aged 18-60yrs, with BMI of 19-31kg/m2.
* Females must be of non-childbearing potential.
* QTc < 450 msec at screening.
* Subjects must be able to give consent and comply with restrictions of study.

Exclusion Criteria:

* Clinically significant CNS, cardiac, pulmonary, metabolic, renal, hepatic or GI condition or history that may place the subject at an unacceptable risk or may interfere with absorption, distribution, metabolism, or excretion of drug.
* Positive urine drug screen.
* Positive urine test for alcohol.
* Positive HIV or Hep B and/or C assay.
* History of regular tobacco use within 3 monts prior to screening or cotinine levels indicative of smoking at screening.
* History of regular alcohol consumption (14 units/week for women and 21 units/week for men).
* History of drug abuse or dependence within 12 months of study.
* Participation in another drug trial within 30 days of first dose.
* Exposure to more than 4 new chemical entities within 12 months of first dose.
* Use of prescription and non-prescription drugs including vitamins, dietary supplements, herbals within 7 days of first dose or St. John's Wort within 28 days of the first dose.
* Consumption of red wine, Seville oranges, grapefruit, or grapefruit juices within 14 days of first dose.
* Donation of blood in excess of 500 mL within 56 days of dosing. No blood donation is allowed 30 days prior to study participation.
* A positive immunochemical fecal occult blood test at screening.
* History of sensitivity to any of the study medications.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of orthostatic hypotension or orthostatic hypotension at screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK580416 doses determined from clinical safety and tolerability data from all adverse event reporting, 12-lead ECGs, vital signs, nursing/physician observation, and safety laboratory tests

SECONDARY OUTCOMES:
Pharmacokinetics of GSK580416 as determined by AUC, Cmax, tmax, half-life, and Ct.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia